CLINICAL TRIAL: NCT05909813
Title: A Feasibility Study on Individualized Piano Instruction (IPI) for Improving Cognition in Breast Cancer Survivors.
Brief Title: Individualized Piano Instruction (IPI) for Improving Cognition in Breast Cancer Survivors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Debbie Anglade, PhD, MSN, RN, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20160725; NCI-2023-00409 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Chemotherapy-Related Cognitive Impairment
MeSH Terms: conditions — Breast Neoplasms; Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized Piano Instruction (IPI) (Experimental): Participants will receive six weeks of individualized piano instruction and two weeks follow-up for a total of eight weeks.
  Interventions: Behavioral: Individualized Piano Keyboard Instruction

INTERVENTIONS:
Behavioral: Individualized Piano Keyboard Instruction — During weeks two through seven, participants will receive a once a week, hour long, in-person individualized piano keyboard instruction as follows:
  1. Warm-up
     1. Scales and Chords: Consisting of scales on seven major keys (C, D, E, F, G, A and B), chord progressions on I, IV, V, I. Two different keys will be learned every week.
     2. 5-finger exercises will be completed four times per week.
  2. Piano Theory and Music
     1. Piano Theory: Playing through Alfred's Basic Adult All-in-One Course, Book 1, to be completed at the ability level of participant, with a least two new pages per lesson.
     2. Chosen Piece: Playing through an instrumental piece chosen by the participant.
  Participants will be asked to practice homework from this lesson daily for 20 minutes per day, until their next weekly lesson.
  Other Names: Individual Piano Instruction; IPI

SUMMARY:
The purpose of this study is to test the study method and procedure for individualized piano instruction (IPI) and its impact on chemotherapy related cognitive impairment (CRCI) symptoms. There have been studies that show the benefits of leaning to play the piano keyboard on cognitive skills in children and elderly populations. The information collected from the program will be used to examine the feasibility of implementing this program permanently

ELIGIBILITY:
Inclusion Criteria:

Patients will be included into the study who:

* Are over 18 years old
* Speaks and read English
* Have been diagnosed and treated for breast cancer (no specific etiology);
* Are experiencing cognitive issues (i.e. actively complain to their physician about struggles with cognitive skills such as memory, attention, executive function, etc.);
* Are 6 months or more out of active treatment;
* Are not currently involved in other brain training programs.

Exclusion Criteria:

* Adults who are diagnosed with a cognitive condition other than CRCI (Such as Alzheimer's, Parkinson's, dementia, Amyotrophic Lateral Sclerosis (ALS), autism, and cerebral palsy.)
* Patients who are in active treatment for breast cancer (Currently hospitalized for chemotherapy or still visiting hospital for outpatient infusion treatment)
* Adults who cannot read and write in English fluently.
* Adults who do not have functional movements in their hands, as assessed by tendon gliding and finger opposition exercises provided by a physical hand therapist.
* Adults who plan to not be in Miami for a period eight weeks or are unable to travel to Sylvester Miami on a weekly basis.
* Adults who are already proficient in piano playing, music theory and play informally or professionally at least once per week.
* Elderly adults, those older than 65 years old.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Post-Individualized Piano Instruction Feasibility Questionnaire | Up to 8 weeks
  An investigator-designed questionnaire will be administered to participants, assessing their opinions about the program. The questionnaire includes multiple sections assessing participant session attendance, the effectiveness of the program, and how enjoyable it was. Total percentage scores will be calculated for each section.
  The Participants' attendance section scores range from "1" to "4" sessions. A higher number of sessions attended indicates greater perceived program feasibility.
  Questions assessing program effectiveness asked participants about their daily and weekly piano routines. Responses range from "not very easily" to "very easily". A higher positive response percentage indicates greater perceived program feasibility.
  Program enjoyment questions asked participants to rate their satisfaction. Responses range from "not enjoyable" to "very enjoyable".A higher positive response percentage indicates greater perceived program feasibility.
Change in Cognition Scores: NIH Toolbox Cognition Battery | Weeks 1, 4 and 8, Up to 8 weeks
  The National Institutes of Health Toolbox Cognition Battery (NIHTB-CB) will be administered to participants to measure change in cognition after individualized piano instruction. The NIHTB-CB consists of tests of multiple constructs, yielding individual test scores and the following summary scores: Total Cognition Composite, Fluid Composite (includes Dimensional Change Card Sort, Flanker Inhibitory Control and Attention, Picture Sequence Memory (Form A), List Sorting Working Memory, and Pattern Comparison tests), and Crystallized Composite (includes Picture Vocabulary and Oral Reading Recognition tests). Scores on the NIHTB-CB will be used to assess severity of chemotherapy-related cognitive injury (CRCI) in participants. Scores range from 59-140, higher scores mean better cognition.
Change in Quality of Life (QOL) Scores: Generalized Anxiety Disorder Assessment (GAD-7) | Weeks 1, 4 and 8, Up to 8 weeks
  The Generalized Anxiety Disorder Assessment (GAD-7) questionnaire will be administered to participants to measure the change in anxiety levels after individualized piano instruction. The GAD-7 consists of seven questions with each possible response scored on a four-point Likert scale ranging from "0" (not at all) to "4" (nearly every day). Higher total scores indicate greater severity of anxiety: 0-4 no to low-risk, 5-9 mild, 10-14 moderate, 15+ severe.
Change in Quality of Life (QOL) Scores: Patient Health Questionnaire (PHQ-9) | Weeks 1, 4 and 8, Up to 8 weeks
  A Patient Health Questionnaire (PHQ-9) will be administered to participants to measure changes in mood after individualized piano instruction. The PHQ-9 consists of nine questions, with each possible response scored on a four-point Likert scale ranging from "0" (not at all) to "3" (nearly every day). Higher total scores indicate greater severity of depression: 0-4 none, 5-9 minimal, 10-14 moderate, 15-19 moderately severe, and 20-27 severe.
Change in Cognition Scores: FACT-Cog | Weeks 1, 4 and 8, Up to 8 weeks
  The Functional Assessment of Cancer Therapy Cognitive Function (FACT-Cog) will be administered to participants to measure change in cognition after individualized piano instruction. The FACT-B is a 33-item questionnaire designed to assess perceived cognitive function and impact on quality of life in cancer patients within four domains: Perceived cognitive impairments, comments from others, perceiving cognitive abilities, and impact on quality of life. Each response within each domain is scored on a five-point Likert scale ranging from "0" (not at all) to 4 (very much). Higher total scores indicate a higher level of cognition and quality of life.
Change in Quality of Life (QOL) Scores: FACT-B | Weeks 1, 4 and 8, Up to 8 weeks
  The Functional Assessment of Cancer Therapy-Breast (FACT-B) will be administered to participants to measure the change in the quality of life after individualized piano instruction (IPI). The FACT-B is a 36-item questionnaire designed to measure five domains of health-related QOL in breast cancer patients: Physical, social, emotional, and functional well-being as well as a breast-cancer subscale (BCS). Each response within each domain is scored on a five-point Likert scale ranging from "0" (not at all) to 4 (very much). Higher scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Anglade, PhD, MSN, RN, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States